CLINICAL TRIAL: NCT00112918
Title: A Randomized, Three Arm Multinational Phase III Study to Investigate Bevacizumab (q3w or q2w) in Combination With Either Intermittent Capecitabine Plus Oxaliplatin (XELOX) (q3w) or Fluorouracil/Leucovorin With Oxaliplatin (FOLFOX-4) Versus FOLFOX-4 Regimen Alone as Adjuvant Chemotherapy in Colon Carcinoma: The AVANT Study
Brief Title: Combination Chemotherapy With or Without Bevacizumab in Treating Patients Who Have Undergone Surgery for High Risk Stage II or Stage III Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000427299; P30CA016042 (NIH); UCLA-0412086-01; ROCHE-BO17920A
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin

ARMS (3):
- FOLFOX4 (Active Comparator): Weeks 1-24: Oxaliplatin was administered as an 85 mg/m^2 intravenous infusion over 2 hours concomitantly with leucovorin as a 200 mg/m^2 infusion over 2 hours, followed by 5-FU, given as a 400 mg/m^2 bolus injection, and then as a 600 mg/m^2 continuous infusion over 22 hours. Leucovorin 200 mg/m^2 (alone), followed by 5-FU 400 mg/m^2 bolus injection, and 5-FU 600 mg/m^2 continuous infusion were repeated on day 2. Cycle length was 2 weeks and cycles were repeated every second week for a total of 12 cycles (24 weeks).
  Weeks 25-48: Observation only.
  Interventions: Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin calcium; Drug: Oxaliplatin
- FOLFOX4 + Bv (Experimental): Weeks 1-24: Bevacizumab 5 mg/kg was administered as an intravenous infusion over 30 - 90 minutes followed by oxaliplatin, administered as an 85 mg/m^2 intravenous infusion over 2 hours (on day 1 only) concomitantly with leucovorin, as a 200 mg/m^2 infusion over 2 hours, followed by 5-FU, given as a 400 mg/m^2 bolus injection, and then as a 600 mg/m^2 continuous infusion over 22 hours. Leucovorin 200 mg/m^2 (alone), followed by 5-FU 400 mg/m^2 bolus injection, and 5-FU 600 mg/m^2 continuous infusion are repeated on day 2. Cycle length is 2 weeks and cycles were repeated every second week for a total of 12 cycles (24 weeks).
  Weeks 25-48: Bevacizumab 7.5 mg/kg was administered as an intravenous infusion over 30 minutes. Cycle length was 3 weeks. Cycles were repeated every 3 weeks for a total of 8 cycles (24 weeks).
  Interventions: Biological: Bevacizumab; Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin calcium; Drug: Oxaliplatin
- XELOX+Bv (Experimental): Weeks 1-24: Bevacizumab 7.5 mg/kg was administered as an intravenous infusion over 30 - 90 minutes followed by oxaliplatin administered as a 130 mg/m^2 intravenous infusion over 2 hours (day 1 every 3 weeks) in combination with capecitabine, which was administered orally at a dose of 1000 mg/m^2 twice daily (equivalent to a total daily dose of 2000 mg/m^2), with first dose the evening of day 1 and last dose the morning of day 15, given as intermittent treatment (3-week cycles consisting of 2 weeks of treatment followed by 1 week without treatment), for a total of 8 cycles (24 weeks).
  Weeks 25-48: Bevacizumab 7.5 mg/kg was administered as an intravenous infusion over 30 minutes. Cycle length was 3 weeks. Cycles were repeated every 3 weeks for a total of 8 cycles (24 weeks).
  Interventions: Biological: Bevacizumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Biological: Bevacizumab — Administered as an intravenous infusion over 30 - 90 minutes.
  Arms: FOLFOX4 + Bv; XELOX+Bv
Drug: Capecitabine — Film-coated tablets
  Other Names: Xeloda®
  Arms: XELOX+Bv
Drug: 5-Fluorouracil (5-FU) — Administered as either a bolus injection or continuous intravenous infusion over 22 hours.
  Arms: FOLFOX4; FOLFOX4 + Bv
Drug: Leucovorin calcium — Administered as a 200 mg/m^2 infusion over 2 hours.
  Arms: FOLFOX4; FOLFOX4 + Bv
Drug: Oxaliplatin — Administered as an intravenous infusion over 2 hours.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab (Bv) may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab after surgery may kill any tumor cells that remain after surgery. It is not yet known whether giving combination chemotherapy together with bevacizumab is more effective than combination chemotherapy alone in treating colon cancer in adjuvant setting.

PURPOSE: This randomized phase III trial is studying two different combination chemotherapy regimens with or without bevacizumab to compare how well they work in treating patients who have undergone surgery for high risk stage II or stage III colon cancer.

DETAILED DESCRIPTION:
This was an open-label Phase III, multicenter, multinational, randomized, 3-arm study designed to evaluate the efficacy and safety of bevacizumab in combination with either intermittent fluorouracil/leucovorin with oxaliplatin (FOLFOX4) or capecitabine plus oxaliplatin (XELOX) versus FOLFOX4 regimen alone, as adjuvant chemotherapy in colon carcinoma.

The treatment phase consisted of two parts of 24 weeks for a total of 48 weeks. The first part (weeks 1 to 24) consisted of treatment with either FOLFOX4, FOLFOX4 in combination with bevacizumab, or XELOX in combination with bevacizumab. The second part (weeks 25 to 48) consisted of single-agent bevacizumab for patients randomized to either bevacizumab-containing arm, but was only an observation period for patients assigned to the FOLFOX4-alone arm.

Patients were to be followed for recurrence/new occurrence of colorectal cancer and survival. Patients who experienced a confirmed recurrence, occurrence of a new colorectal cancer during therapy, or experienced unacceptable toxicity were to be taken off study treatment but remain in study follow-up. Patients that came off therapy due to a confirmed recurrence/appearance of new colorectal cancer, were to be followed for survival until the end of the study follow-up period. The primary analysis was performed 36 months after the last patient has been randomized. After the primary analysis, patients continue to be followed for survival for at least a further 2 years ie, until all patients have been followed-up for at least 5 years following randomization.

ELIGIBILITY:
Inclusion Criteria

1. Signed written informed consent obtained prior to any study specific screening procedures.
2. Patient willing and able to comply with the protocol.
3. Age ≥ 18 years-of-age.
4. Histologically confirmed colon carcinoma, American Joint Cancer Committee/Union Internationale Contre le Cancer (AJCC/UICC) Stage II or Stage III defined as a tumor location ≥ 15 cm from the anal verge by endoscopy or above the peritoneal reflection at surgery. The patient was not to be a candidate for (neo) adjuvant radiotherapy. Note: Stage II patients were to be considered as high-risk patients fulfilling one of the following criteria:

   * T4 tumours,
   * Patients presenting with bowel obstruction or perforation,
   * Histological signs of vascular invasion (i.e. blood and lymphatic vessels) or perineural invasion,
   * Patients aged less than 50 years,
   * Patients with sub-optimal surgery (less than 12 nodes analyzed).
5. Curative surgery not less than 4 and not more than 8 weeks prior to randomization.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Life expectancy of ≥ 5 years.

Exclusion Criteria

1. Macroscopic or microscopic evidence of remaining tumour. Patients should never have had any evidence of metastatic disease (including presence of tumour cells in the ascites). The isolated finding of cytokeratin positive cells in bone marrow is not considered evidence of metastatic disease for purposes of this study.
2. Carcinoembryonic antigen > 1.5 x upper limit of normal (ULN) after surgery (during screening period).
3. For patients with colostomy, unwilling to delay revision until at least 28 days after treatment completion.
4. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, not fully healed wounds, or anticipation of the need for major surgical procedure during the course of the study. Any central venous access device (CVAD) for chemotherapy administration must be inserted at least 2 days prior to treatment start.
5. Previous anti-angiogenic treatment for any malignancy; cytotoxic chemotherapy, radiotherapy or immunotherapy for colon cancer.
6. Other malignancies within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix).
7. Females with a positive or no pregnancy test (within 7 days before treatment start) unless childbearing potential can be otherwise excluded (postmenopausal i.e. amenorrheic for at least 2 years, hysterectomy or oophorectomy).
8. Lactating women.
9. Fertile women (< 2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception.
10. History or evidence upon physical examination of central nervous disease (CNS) disease (eg, primary brain tumour, seizure not controlled with standard medical therapy, any brain metastases).
11. History of psychiatric disability judged by the investigator to be clinically significant, precluding informed consent or interfering with compliance for oral drug intake.
12. Clinically significant (ie, active) cardiovascular disease. This includes, but is not limited to, the following examples: cerebrovascular accidents (≤ 6 months prior to randomization), myocardial infarction (≤ 1 year prior to randomization), uncontrolled hypertension (>150/100 mmHg) while receiving chronic medication, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, clinically significant electrocardiogram (ECG) findings (e.g. QTc ≥ 440 msecs [male] 460 msecs [female] or ≥ 2º atrioventricular block, etc.).

    Patients who suffer from serious cardiac arrhythmia requiring medication can enter the study only if they are considered to be in a stable condition regarding both the arrhythmia and their medication. Patients with pacemakers are allowed to enter the study only if they are considered as being in a stable condition. In case of doubt, the investigator should obtain a consultation with a local cardiologist.
13. Lack of physical integrity of the upper gastro-intestinal tract, malabsorption syndrome, or inability to take oral medication.
14. Interstitial pneumonia or extensive symptomatic fibrosis of the lungs.
15. Known peripheral neuropathy ≥ Common terminology criteria for adverse events (CTCAE) version 3.0 Grade 1. Absence of deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible.
16. Organ allografts requiring immunosuppressive therapy.
17. Serious, non-healing wound, ulcer, or bone fracture.
18. Evidence of bleeding diathesis or coagulopathy.
19. Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes.
20. Chronic, daily treatment with high-dose aspirin (> 325 mg/day) or clopidogrel (> 75 mg/day).
21. Chronic treatment with corticosteroids (dose of ≥ 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids).
22. Serious intercurrent infections (uncontrolled or requiring treatment).
23. Known dihydropyrimidine dehydrogenase deficiency.
24. Current or recent (within the 28 days prior to randomization) treatment with another investigational drug or participation in another investigational study.
25. Patients with known allergy to Chinese hamster ovary cell proteins or other recombinant human or humanized antibodies or to any excipients of bevacizumab formulation, platinum compounds or to any other components of the study drugs.
26. History or presence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or patient at high risk from treatment complications.
27. Presence of proteinuria at baseline as defined by:

    - Patients with > 1 g of protein/24 hour by a 24-hour urine collection.
28. Any laboratory values at baseline are as follows:

Haematology:

* Absolute neutrophil count (ANC) < 1.5 x 109/L
* Platelet count < 100 x 10^9/L
* Haemoglobin < 9 g/dL (may be transfused to maintain or exceed this level)
* International normalized ratio (INR) > 1.5
* Activated partial prothrombin time (APTT) ≥ 1.5 x ULN

Biochemistry:

* Total bilirubin > 1.5 x ULN
* aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT) > 2.5 x ULN
* Alkaline phosphatase (ALP) > 2.5 x ULN
* Serum creatinine > 1.5 x ULN or creatinine clearance ≤ 50 mL/min (e.g. Cockcroft-Gault formula).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3451 (Actual)
Dates: Start 2004-12; Primary Completion 2010-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Randolph Hecht, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Cohen R, Taieb J, Fiskum J, Yothers G, Goldberg R, Yoshino T, Alberts S, Allegra C, de Gramont A, Seitz JF, O'Connell M, Haller D, Wolmark N, Erlichman C, Zaniboni A, Lonardi S, Kerr R, Grothey A, Sinicrope FA, Andre T, Shi Q. Microsatellite Instability in Patients With Stage III Colon Cancer Receiving Fluoropyrimidine With or Without Oxaliplatin: An ACCENT Pooled Analysis of 12 Adjuvant Trials. J Clin Oncol. 2021 Feb 20;39(6):642-651. doi: 10.1200/JCO.20.01600. Epub 2020 Dec 23. PMID 33356421
- [Derived] Chibaudel B, Henriques J, Rakez M, Brenner B, Kim TW, Martinez-Villacampa M, Gallego-Plazas J, Cervantes A, Shim K, Jonker D, Guerin-Meyer V, Mineur L, Banzi C, Dewdney A, Dejthevaporn T, Bloemendal HJ, Roth A, Moehler M, Aranda E, Van Cutsem E, Tabernero J, Schmoll HJ, Hoff PM, Andre T, de Gramont A. Association of Bevacizumab Plus Oxaliplatin-Based Chemotherapy With Disease-Free Survival and Overall Survival in Patients With Stage II Colon Cancer: A Secondary Analysis of the AVANT Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2020425. doi: 10.1001/jamanetworkopen.2020.20425. PMID 33074326
- [Derived] Salem ME, Yin J, Goldberg RM, Pederson LD, Wolmark N, Alberts SR, Taieb J, Marshall JL, Lonardi S, Yoshino T, Kerr RS, Yothers G, Grothey A, Andre T, De Gramont A, Shi Q. Evaluation of the change of outcomes over a 10-year period in patients with stage III colon cancer: pooled analysis of 6501 patients treated with fluorouracil, leucovorin, and oxaliplatin in the ACCENT database. Ann Oncol. 2020 Apr;31(4):480-486. doi: 10.1016/j.annonc.2019.12.007. Epub 2020 Jan 16. PMID 32085892
- [Derived] Andre T, Vernerey D, Im SA, Bodoky G, Buzzoni R, Reingold S, Rivera F, McKendrick J, Scheithauer W, Ravit G, Fountzilas G, Yong WP, Isaacs R, Osterlund P, Liang JT, Creemers GJ, Rakez M, Van Cutsem E, Cunningham D, Tabernero J, de Gramont A. Bevacizumab as adjuvant treatment of colon cancer: updated results from the S-AVANT phase III study by the GERCOR Group. Ann Oncol. 2020 Feb;31(2):246-256. doi: 10.1016/j.annonc.2019.12.006. Epub 2019 Dec 18. PMID 31959341
- [Derived] Taieb J, Shi Q, Pederson L, Alberts S, Wolmark N, Van Cutsem E, de Gramont A, Kerr R, Grothey A, Lonardi S, Yoshino T, Yothers G, Sinicrope FA, Zaanan A, Andre T. Prognosis of microsatellite instability and/or mismatch repair deficiency stage III colon cancer patients after disease recurrence following adjuvant treatment: results of an ACCENT pooled analysis of seven studies. Ann Oncol. 2019 Sep 1;30(9):1466-1471. doi: 10.1093/annonc/mdz208. PMID 31268130
- [Derived] de Gramont A, Van Cutsem E, Schmoll HJ, Tabernero J, Clarke S, Moore MJ, Cunningham D, Cartwright TH, Hecht JR, Rivera F, Im SA, Bodoky G, Salazar R, Maindrault-Goebel F, Shacham-Shmueli E, Bajetta E, Makrutzki M, Shang A, Andre T, Hoff PM. Bevacizumab plus oxaliplatin-based chemotherapy as adjuvant treatment for colon cancer (AVANT): a phase 3 randomised controlled trial. Lancet Oncol. 2012 Dec;13(12):1225-33. doi: 10.1016/S1470-2045(12)70509-0. Epub 2012 Nov 16. PMID 23168362

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was stratified according to geographic region and disease stage (high-risk stage II or stage III N1 or stage III N2). The primary analysis population consisted of patients with Stage III disease.
Groups:
- FOLFOX4: Weeks 1-24: Oxaliplatin was administered as an 85 mg/m^2 intravenous infusion over 2 hours concomitantly with leucovorin as a 200 mg/m^2 infusion over 2 hours, followed by 5-fluorouracil (5-FU), given as a 400 mg/m^2 bolus injection, and then as a 600 mg/m^2 continuous infusion over 22 hours. Leucovorin 200 mg/m^2 (alone), followed by 5-FU 400 mg/m^2 bolus injection, and 5-FU 600 mg/m^2 continuous infusion were repeated on day 2. Cycle length was 2 weeks and cycles were repeated every second week for a total of 12 cycles (24 weeks).
  Weeks 25-48: Observation only.
Period: Overall Study
Arm/Group | FOLFOX4 | FOLFOX4 + Bv | XELOX+Bv
Started | 1151 | 1155 | 1145
Received Treatment | 1126 | 1145 (Includes two patients from FOLFOX4 who received Bv and were assigned to FOLFOX4+Bv safety analysis) | 1135
Stage III Disease Population | 955 | 960 | 952
Completed | 854 (Represents patients alive in follow-up at the time of final data cut-off (30 June 2012)) | 810 (Represents patients alive in follow-up at the time of final data cut-off (30 June 2012)) | 846 (Represents patients alive in follow-up at the time of final data cut-off (30 June 2012))
Not Completed | 297 | 345 | 299

BASELINE CHARACTERISTICS:
Population: Baseline Measures are based on the Intent-to-Treat - Stage III Disease Patient Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFOX4 | FOLFOX4 + Bv | XELOX+Bv | Total
Number analyzed (Participants) | 955 | 960 | 952 | 2867
Age, Customized [Number; unit: participants]
  <40 | 77 | 74 | 68 | 219
  40-65 | 603 | 625 | 588 | 1816
  >=65 | 275 | 261 | 296 | 832
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 425 | 473 | 432 | 1330
  Male | 530 | 487 | 520 | 1537
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 139 | 115 | 123 | 377
  Black or African American | 6 | 13 | 14 | 33
  White | 791 | 813 | 795 | 2399
  Other | 18 | 18 | 20 | 56

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival in Stage III Cancer Patients - Time to Event
Description: Disease-free survival (DFS) was defined as the time from the date of randomization to the time of a recurrence, a new occurrence of colorectal cancer or death due to any cause, whichever occurred first. Patients without an event were censored at the last date the patient was known to be disease-free. Recurrence and new occurrence of colorectal cancer were based on tumor assessments made by the investigator. Patients with no tumor assessments after baseline but still alive at the time of the clinical cut-off were censored at day 1.
Time Frame: From first patient randomized until the data cut-off date of 30 June 2010 (36 months after the last patient randomized).
Population: The primary population for efficacy analyses was the intent to treat population (ITT; all randomized patients) with stage III disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOX4 | FOLFOX4 + Bv | XELOX+Bv
Number analyzed (Participants) | 955 | 960 | 952
months | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to the low number of events. | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to the low number of events. | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to the low number of events.
Statistical Analysis 1: Comparison: FOLFOX4 vs FOLFOX4 + Bv vs XELOX+Bv; Adjustments for multiplicity was done using a closed test procedure which tests for differences between all three treatment groups at the 5% alpha level first. Only in case of a significant result, the pair-wise comparison between the control arm and each of the bevacizumab arm will be tested, again at the 5% alpha level; Test type: Superiority or Other; p = 0.2024, Closed test procedure

2. Secondary Outcome: Overall Survival in Stage III Cancer Patients - Time to Event
Description: Overall survival was defined as the time between date of randomization and date of death due to any cause. Patients not reported as having died at the time of the analysis were censored at the date they were last known to be alive.
Time Frame: From first patient randomized until the clinical data cut-off date of 30 June 2010 (36 months after the last patient randomized).
Population: ITT patients with Stage III disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOX4 | FOLFOX4 + Bv | XELOX+Bv
Number analyzed (Participants) | 955 | 960 | 952
months | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to the low number of events. | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to the low number of events. | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to the low number of events.

3. Primary Outcome: Disease-free Survival in Stage III Cancer Patients - Number of Events
Description: A disease-free survival (DFS) event was composed of a recurrence, a new occurrence of colorectal cancer or death due to any cause. Recurrence and new occurrence of colorectal cancer were based on tumor assessments made by the investigator. Triggering events for DFS are reported; a patient can have both recurrence and a new occurrence of colon cancer.
Time Frame: From first patient randomized until the data cut-off date of 30 June 2010 (36 months after the last patient randomized).
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | FOLFOX4 | FOLFOX4 + Bv | XELOX+Bv
Number analyzed (Participants) | 955 | 960 | 952
participants
  Patients with a DFS event | 237 | 280 | 253
  Recurrence | 219 | 253 | 223
  New Occurrence | 3 | 8 | 6
  Death | 17 | 21 | 25
  Patients without events | 718 | 680 | 699

4. Secondary Outcome: Overall Survival in Stage III Cancer Patients - Number of Events
Description: An overall survival event was death due to any cause.
Time Frame: as for outcome 2
Population: ITT patients with Stage III disease.
Measure: Number; unit: participants
Arm/Group | FOLFOX4 | FOLFOX4 + Bv | XELOX+Bv
Number analyzed (Participants) | 955 | 960 | 952
participants
  Patients with events | 115 | 151 | 145
  Patients without events | 840 | 809 | 807

5. Secondary Outcome: Overall Survival in Stage III Cancer Patients - Time to Event: Final Analysis
Description: Overall survival was defined as the time between date of randomization and date of death due to any cause. Patients not reported as having died at the time of the clinical cut-off date (30 June 2012) were censored at the date they were last known to be alive.
Time Frame: From first patient randomized until the final data cut-off date of 30 June 2012 (5 years after the last patient randomized).
Population: ITT patients with Stage III disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFOX4 | FOLFOX4 + Bv | XELOX+Bv
Number analyzed (Participants) | 955 | 960 | 952
months | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to the low number of events. | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to the low number of events. | NA [NA to NA] — Median time to event and 95% confidence intervals could not be estimated due to the low number of events.

6. Secondary Outcome: Overall Survival in Stage III Cancer Patients - Number of Events: Final Analysis
Description: An overall survival event was death due to any cause.
Time Frame: as for outcome 5
Population: ITT patients with Stage III disease.
Measure: Number; unit: participants
Arm/Group | FOLFOX4 | FOLFOX4 + Bv | XELOX+Bv
Number analyzed (Participants) | 955 | 960 | 952
participants
  Patients with events | 161 | 202 | 182
  Patients without events | 794 | 758 | 770

ADVERSE EVENTS:
Time Frame: All adverse events occurring between the date of first drug intake and 28 days after last drug intake, regardless of which treatment group the patient was randomized to.
Arm/Group | FOLFOX4 | FOLFOX4 + Bv | XELOX+Bv
Serious Adverse Events (participants affected / at risk) | 226/1126 | 297/1145 | 284/1135
Other Adverse Events (participants affected / at risk) | 1112/1126 | 1127/1145 | 1117/1135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX4 (N=1126) | FOLFOX4 + Bv (N=1145) | XELOX+Bv (N=1135)
Diarrhoea (Gastrointestinal disorders) | 28 | 28 | 62
Abdominal pain (Gastrointestinal disorders) | 11 | 14 | 18
Vomiting (Gastrointestinal disorders) | 7 | 11 | 16
Intestinal obstruction (Gastrointestinal disorders) | 6 | 9 | 7
Nausea (Gastrointestinal disorders) | 0 | 4 | 7
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 7 | 3
Enteritis (Gastrointestinal disorders) | 3 | 0 | 5
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 4 | 2
Subileus (Gastrointestinal disorders) | 1 | 4 | 2
Colitis (Gastrointestinal disorders) | 0 | 1 | 5
Abdominal adhesions (Gastrointestinal disorders) | 2 | 0 | 2
Gastritis (Gastrointestinal disorders) | 3 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 2 | 2
Small intestinal perforation (Gastrointestinal disorders) | 0 | 4 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 2 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 2 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1 | 0
Caecitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal angina (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal dilatation (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal prolapse (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal strangulation (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1 | 0
Device related infection (Infections and infestations) | 8 | 12 | 4
Pneumonia (Infections and infestations) | 3 | 4 | 5
Urinary tract infection (Infections and infestations) | 2 | 5 | 4
Sepsis (Infections and infestations) | 4 | 3 | 3
Gastroenteritis (Infections and infestations) | 1 | 5 | 3
Infection (Infections and infestations) | 5 | 3 | 1
Abdominal abscess (Infections and infestations) | 2 | 4 | 2
Catheter site infection (Infections and infestations) | 4 | 4 | 0
Neutropenic sepsis (Infections and infestations) | 4 | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 2 | 0
Anal abscess (Infections and infestations) | 0 | 3 | 1
Cellulitis (Infections and infestations) | 3 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 2 | 1
Device related sepsis (Infections and infestations) | 1 | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 2
Abscess (Infections and infestations) | 0 | 2 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Neutropenic infection (Infections and infestations) | 1 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 2 | 0
Septic shock (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Aspergillosis (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 | 0
Candida sepsis (Infections and infestations) | 0 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Enteritis infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0 | 0
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0 | 0
Incision site cellulitis (Infections and infestations) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 1
Intestinal fistual infection (Infections and infestations) | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1
Overgrowth bacterial (Infections and infestations) | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 1 | 0
Puncture site infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1 | 0
Wound abscess (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 9 | 16 | 12
Hypertension (Vascular disorders) | 1 | 2 | 13
Venous thrombosis (Vascular disorders) | 3 | 5 | 1
Jugular vein thrombosis (Vascular disorders) | 2 | 3 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 2 | 2
Venous thrombosis limb (Vascular disorders) | 0 | 3 | 2
Hypertensive crisis (Vascular disorders) | 0 | 3 | 1
Hypotension (Vascular disorders) | 0 | 2 | 1
Thrombophlebitis (Vascular disorders) | 1 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0
Arterial stenosis (Vascular disorders) | 0 | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 1
Axillary vein thrombosis (Vascular disorders) | 0 | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 20 | 10 | 16
Non-cardiac chest pain (General disorders) | 1 | 2 | 5
Sudden death (General disorders) | 0 | 2 | 3
Asthenia (General disorders) | 0 | 3 | 1
Chest pain (General disorders) | 1 | 2 | 1
Extravasation (General disorders) | 0 | 0 | 2
Medical device complication (General disorders) | 1 | 1 | 0
Multi-organ failure (General disorders) | 2 | 0 | 0
Thrombosis in device (General disorders) | 1 | 0 | 1
Adhesion (General disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0
Device leakage (General disorders) | 1 | 0 | 0
Device malfunction (General disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Hernia obstructive (General disorders) | 0 | 0 | 1
Hyperpyrexia (General disorders) | 1 | 0 | 0
Infusion site thrombosis (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 0 | 1
Visceral pain (General disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 18 | 18 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 9 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Idiopathic thrombocytopenia purpura (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 15 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 10 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 5 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 3 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1
Convulsion (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Leukoaraiosis (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 0 | 1
Neurotoxicity (Nervous system disorders) | 1 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 5 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 4
Coronary artery disease (Cardiac disorders) | 1 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 2
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Arteriospasm coronary (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Cardiac asthma (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Paroxysmal arrhythmia (Cardiac disorders) | 0 | 0 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 2 | 2
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2
Accident at work (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 5 | 3 | 1
Hypersensitivity (Immune system disorders) | 3 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 3 | 0
Anaphylactic shock (Immune system disorders) | 2 | 0 | 1
Anaphylactiod reaction (Immune system disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 2
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 2 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0
Nephrogenic diabetes insipidus (Renal and urinary disorders) | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood glucose fluctuation (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar-Plantar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1
Alcoholism (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0
Pregnancy of partner (Social circumstances) | 0 | 1 | 0
Central venous catheter removal (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFOX4 (N=1126) | FOLFOX4 + Bv (N=1145) | XELOX+Bv (N=1135)
Nausea (Gastrointestinal disorders) | 725 | 761 | 720
Diarrhoea (Gastrointestinal disorders) | 620 | 699 | 699
Vomiting (Gastrointestinal disorders) | 385 | 394 | 460
Stomatitis (Gastrointestinal disorders) | 310 | 360 | 246
Constipation (Gastrointestinal disorders) | 308 | 324 | 219
Abdominal pain (Gastrointestinal disorders) | 220 | 227 | 214
Dyspepsia (Gastrointestinal disorders) | 126 | 162 | 84
Abdominal pain upper (Gastrointestinal disorders) | 86 | 118 | 113
Haemorrhoids (Gastrointestinal disorders) | 29 | 68 | 41
Peripheral sensory neuropathy (Nervous system disorders) | 430 | 430 | 436
Paraesthesia (Nervous system disorders) | 310 | 328 | 314
Neuropathy peripheral (Nervous system disorders) | 252 | 234 | 204
Headache (Nervous system disorders) | 169 | 284 | 219
Dysgeusia (Nervous system disorders) | 237 | 222 | 152
Dysaesthesia (Nervous system disorders) | 128 | 106 | 128
Dizziness (Nervous system disorders) | 102 | 117 | 79
Neurotoxicity (Nervous system disorders) | 60 | 69 | 50
Lethargy (Nervous system disorders) | 44 | 50 | 59
Fatigue (General disorders) | 404 | 425 | 355
Asthenia (General disorders) | 241 | 251 | 250
Pyrexia (General disorders) | 186 | 185 | 106
Mucosal inflammation (General disorders) | 85 | 85 | 57
Temperature intolerance (General disorders) | 61 | 61 | 50
Oedema peripheral (General disorders) | 54 | 62 | 45
Neutropenia (Blood and lymphatic system disorders) | 660 | 567 | 273
Thrombocytopenia (Blood and lymphatic system disorders) | 331 | 115 | 99
Anaemia (Blood and lymphatic system disorders) | 116 | 89 | 74
Leukopenia (Blood and lymphatic system disorders) | 79 | 55 | 34
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 98 | 119 | 435
Alopecia (Skin and subcutaneous tissue disorders) | 231 | 241 | 73
Rash (Skin and subcutaneous tissue disorders) | 114 | 112 | 110
Dry skin (Skin and subcutaneous tissue disorders) | 52 | 66 | 50
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 65 | 28
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 228 | 424 | 216
Cough (Respiratory, thoracic and mediastinal disorders) | 86 | 120 | 41
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 57 | 74 | 73
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 17 | 91 | 74
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 37 | 28 | 79
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 52 | 59 | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 | 140 | 122
Pain in extremity (Musculoskeletal and connective tissue disorders) | 63 | 78 | 116
Back pain (Musculoskeletal and connective tissue disorders) | 79 | 87 | 66
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 35 | 86 | 46
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 70 | 56
Hypertension (Vascular disorders) | 196 | 472 | 468
Decreased appetite (Metabolism and nutrition disorders) | 268 | 324 | 295
Insomnia (Psychiatric disorders) | 135 | 132 | 91
Anxiety (Psychiatric disorders) | 45 | 60 | 61
Nasopharyngitis (Infections and infestations) | 76 | 92 | 70
Upper respiratory tract infection (Infections and infestations) | 52 | 87 | 55
Weight increased (Investigations) | 58 | 81 | 68
Weight decreased (Investigations) | 26 | 56 | 61
Lacrimation increased (Eye disorders) | 70 | 69 | 35
Drug hypersensitivity (Immune system disorders) | 66 | 72 | 32
Proteinuria (Renal and urinary disorders) | 19 | 73 | 69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.